CLINICAL TRIAL: NCT04114734
Title: Park Rx, Physical Activity and Other Health Benefits Among Low-income Children
Brief Title: Park Rx and Physical Activity Among Low-income Children
Acronym: ParkRx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: Unity Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL147574 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-10-03 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Physical Activity; Mental Health Wellness 1
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to get Park Rx or to receive care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Park Rx (Experimental): Participants will be given a park prescription as part of their treatment plan
  Interventions: Behavioral: Park Rx
- No Park Rx (No Intervention): Usual care only

INTERVENTIONS:
Behavioral: Park Rx — Participants will be advised to visit a specific park at a specific frequency and duration
  Arms: Park Rx

SUMMARY:
This study is a randomized controlled trial to evaluate ParkRx, a clinic-based counseling intervention in which health care providers prescribe park visits at a specific frequency, duration, and includes instructions for physical activity in the parks. We will assess whether prescribing visits to specific parks changes physical activity levels and improves health and mental health outcomes among low-income pediatric patients.

DETAILED DESCRIPTION:
Park prescriptions are formal clinical encouragements for patients to engage in more physical activity outdoors. From the beginning, ParkRx has been perceived as a common-sense solution to physical inactivity and to increasing the time children might be spending outdoors in nature. In spite of a lack of rigorous evidence that it is effective, the ParkRx concept is currently being widely disseminated and has been embraced by multiple national organizations. Unity Health, a federally qualified community health center in Washington, DC, is currently implementing park prescriptions for its largely low-income and minority population, a group at high risk of chronic diseases, physical inactivity and obesity. In partnership with Unity Health, we propose to conduct a randomized controlled trial (RCT) to prospectively evaluate Park Rx's impact on physical activity, as well as other secondary health outcomes in pediatric patients. Our specific aims are: 1) to test whether Park Rx will increase park visits and accelerometry-measured physical activity among children; 2) to identify any biological impacts of Park Rx on health, including impact on hypercholesterolemia, hypertriglyceridemia, HbA1C, overweight and obesity, for those patients with relevant diagnoses; 3) to explore impacts on mental health, including stress and measures of cognitive functioning; and 4) to determine whether there are age and gender differences in adherence to and impact of Park Rx. The results of this study will quantify the effectiveness of Park Rx and inform its future dissemination.

ELIGIBILITY:
Inclusion Criteria:

* ages >6 and <16 with one or more diagnoses of chronic conditions that usually require two or more routine health care provider visits per year.
* ADHD, or
* Overweight or obesity, or
* hypertriglyceridemia or
* hypercholesterolemia, or
* pre-diabetes or
* Type 2 diabetes. AND
* Likely to live in the Washington DC area in the next 2 years.

Exclusion Criteria:

- Individuals who have previously been given a park prescription

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity | Baseline, 3 months, 6 months 12 months and 2 years
  Accelerometer measured

SECONDARY OUTCOMES:
Change in Cognition | Baseline, 3 months, 6 months 12 months and 2 years
  We will use the NIH toolbox A)The Flanker Inhibitory Control Test; B) Dimensional Change Card Sort Test C) List Sorting Working Memory Test

OTHER OUTCOMES:
Change in BMI percentile | 2 years
  We will review the electronic health record for BMI
Change in Lipids | 2 years
  EHR review

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Cohen, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed we will de-identify data and post on the ICSPR website
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At study completion
Access Criteria: not yet available

REFERENCES:
- [Derived] Cohen DA, Zarr RL, Estrada EL, Zhong H, Han B. The Park RX RCT: Impact on Physical Activity Among Youth. Am J Prev Med. 2025 Oct 14;70(3):108154. doi: 10.1016/j.amepre.2025.108154. Online ahead of print. PMID 41101405
- [Derived] Cohen DA, Zarr R, Estrada E, Zhong H, Han B. Association of children's electronic media use with physical activity, cognitive function, and stress. Prev Med. 2025 Jan;190:108184. doi: 10.1016/j.ypmed.2024.108184. Epub 2024 Nov 26. PMID 39592015
- [Derived] Zarr R, Han B, Estrada E, Cohen DA. The Park Rx trial to increase physical activity among low-income youth. Contemp Clin Trials. 2022 Nov;122:106930. doi: 10.1016/j.cct.2022.106930. Epub 2022 Sep 19. PMID 36184966